CLINICAL TRIAL: NCT07400107
Title: Efficacy and Safety of NNC0487-0111 s.c. Once-weekly Compared to Semaglutide s.c. Once-weekly in Participants With Overweight or Obesity, and Type 2 Diabetes (AMAZE 8)
Brief Title: AMAZE 8: A Research Study Investigating How Well the Medicine NNC0487-0111 Compared to Semaglutide Helps People With Excess Body Weight and Type 2 Diabetes Lose Weight
Acronym: AMAZE 8
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9490-8028; U1111-1313-8017 (Other: World Health Organization (WHO)); 2024-520446-31 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0487-0111 (Experimental): Participants will receive NNC0487-0111 and placebo matched to semaglutide subcutaneously once weekly as an adjunct to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: NNC0487-0111; Drug: Placebo (matched to semaglutide)
- Semaglutide (Active Comparator): Participants will receive semaglutide and placebo matched to NNC0487-0111 subcutaneously once weekly as an adjunct to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Semaglutide; Drug: Placebo (matched to NNC0487-0111)

INTERVENTIONS:
Drug: NNC0487-0111 — NNC0487-0111 will be administered subcutaneously using PDS290 pre-filled pen-injectors to one of the body parts: thigh, abdomen or upper arm.
  Arms: NNC0487-0111
Drug: Semaglutide — Semaglutide will be administered subcutaneously using PDS290 pre-filled pen-injectors to one of the body parts: thigh, abdomen or upper arm.
  Arms: Semaglutide
Drug: Placebo (matched to NNC0487-0111) — Placebo matched to NNC0487-0111 will be administered subcutaneously using pre- filled pen-injectors to one of the body parts: thigh, abdomen or upper arm.
  Arms: Semaglutide
Drug: Placebo (matched to semaglutide) — Placebo matched to semaglutide will be administered subcutaneously using pre-filled pen-injectors to one of the body parts: thigh, abdomen or upper arm.
  Arms: NNC0487-0111

SUMMARY:
The purpose of this clinical study is to find out if NNC0487-0111 is safe and effective for treating people who have excess body weight and type 2 diabetes. Participant will receive 2 injections every week: an active medicine and a placebo, both taken as injections under the skin once a week. The placebo is a treatment with no active medicine in it and will be given to all participants. In addition to placebo, participants will receive either of the active medicine NNC0487-0111 (the treatment being tested) or Semaglutide (an approved and commonly prescribed treatment used as comparator). Which treatment participants get is decided by chance.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female (sex at birth).
* Age 18 years or above at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus ≥ 180 days before screening.
* Haemoglobin A1c (HbA1c) 7-10 percentage (%) (53-86 millimole per mole [mmol/mol]) (both inclusive) as measured by the central laboratory at screening.
* Treatment with lifestyle intervention, and/or 0-3 marketed oral antidiabetic drugs (OAD)s (metformin, α-glucosidase inhibitors (AGI), glinides, sodium-glucose cotransporter 2 inhibitor (SGLT2i), thiazolidinediones, or sulfonylureas (SU) as a single agent or in combination) according to local label. Treatment with oral antidiabetic drugs should be stable (same drug(s), dose and dosing frequency) before screening.

Key Exclusion Criteria:

* Renal impairment with estimated Glomerular Filtration Rate (eGFR) < 30 milliliter (mL)/ minute (min)/1.73 meter squared (m^2) (2021 Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula), at screening.
* Participant with diabetic retinopathy or maculopathy who received treatment with retinal photocoagulation, vitrectomy or anti-Vascular Endothelial Growth Factor (anti-VEGF) within 180 days before screening or are expected to require treatment within 180 days after screening. Diabetic retinopathy or maculopathy must be verified by an eye examination performed within 90 days before screening or in the period between screening and randomization. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire question 8.
* Recurrent severe hypoglycaemic episodes within the last year as judged by the investigator.
* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonists (RA), dual GLP-1/gastric inhibitory peptide (GIP) RAs (or any other GLP-1 based treatment), or amylin analogues before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-05-20 (Estimated); Primary Completion 2028-12-12 (Estimated); Study Completion 2029-01-26 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to week 84
  Measured as percentage of body weight.

SECONDARY OUTCOMES:
Change in waist circumference | From baseline (week 0) to week 84
  Measured as centimeter (cm).
Change in systolic blood pressure (SBP) | From baseline (week 0) to week 84
  Measured as millimeter of mercury (mmHg).
Change in body weight | From baseline (week 0) to week 84 and week 104
  Measured as kilograms (kg).
Change in body mass index (BMI) | From baseline (week 0) to week 84 and week 104
  Measured as kilograms per meter squared (kg/m^2).
Number of participants with achievement of in haemoglobin A1c (HbA1c) < 7.0 percent (%) (yes/no) | From baseline (week 0) to week 84
  Measured as count of participants.
Number of participants with achievement of HbA1c ≤ 6.5% (yes/no) | From baseline (week 0) to week 84
  Measured as count of participants.
Number of participants with achievement of HbA1c < 5.7% (yes/no) | From baseline (week 0) to week 84
  Measured as count of participants.
Change in fasting plasma glucose (FPG) measured as millimole per liter (mmol/L) | From baseline (week 0) to week 84
  Measured as mmol/L.
Change in FPG measured as milligrams per deciliter (mg/dL) | From baseline (week 0) to week 84
  Measured as mg/dL.
Ratio to baseline: change in fasting insulin | From baseline (week 0) to week 84
  Measured as ratio.
Ratio to baseline: change in urinary albumin-to-creatinine ratio (UACR) | From baseline (week 0) to week 84
  Measured as ratio.
Change in diastolic blood pressure (DBP) | From baseline (week 0) to week 84
  Measured as mmHg.
Ratio to baseline: change in total cholesterol | From baseline (week 0) to week 84
  Measured as ratio.
Ratio to baseline: change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to week 84
  Measured as ratio.
Ratio to baseline: change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to week 84
  Measured as ratio.
Ratio to baseline: change in very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to week 84
  Measured as ratio.
Ratio to baseline: change in non-HDL cholesterol | From baseline (week 0) to week 84
  Measured as ratio.
Ratio to baseline: change in triglycerides | From baseline (week 0) to week 84
  Measured as ratio.
Ratio to baseline: change in high-sensitivity C-reactive protein (hsCRP) | From baseline (week 0) to week 84
  Measured as ratio.
Number of Treatment Emergent Adverse Events (TEAEs) | From baseline (week 0) to week 84 and week 109
  Measured as events.
Number of Treatment Emergent Serious Adverse Events (TESAEs) | From baseline (week 0) to week 84 and week 109
  Measured as events.
Number of TEAEs leading to permanent treatment discontinuation | From baseline (week 0) to week 84 and week 109
  Measured as events.
Number of treatment-emergent clinically significant hypoglycaemic episodes (level 2) (< 3.0 millimole per liter [mmol/L] (54 milligrams per deciliter [mg/dL]), confirmed by a blood glucose (BG) meter) | From baseline (week 0) to week 84 and week 109
  Measured as episodes.
Number of treatment-emergent severe hypoglycaemic episodes (level 3): hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold | From baseline (week 0) to week 84 and week 109
  Measured as episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (119):
- United States (10):
  - Encore Medical Research LLC, Hollywood, Florida
  - Optimal Research Sites, Orange City, Florida
  - Encore Medical Research of Weston, Weston, Florida
  - Endocrine Research Solutions, Inc, Roswell, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Endo And Metab Cons, Rockville, Maryland
  - Arcturus Healthcare, PLC., Troy, Michigan
  - Velocity Clin Res, Dallas, Dallas, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Selma Medical Associates, Winchester, Virginia
- Argentina (3):
  - Centro de Investigaciones Metabólicas, Capital Federal, Buenos Aires
  - Centro Médico CIMEL, Lanús Este, Buenos Aires
  - Centro Médico Privado San Vicente Diabetes, Córdoba
- Brazil (4):
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - i9 Pesquisas Clínicas, Campinas, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - BR Trials - Ensaios Clínicos e Consultoria Ltda., São Paulo, São Paulo
- Bulgaria (10):
  - Dr. Tatyana Metalova - AIPSMCE EOOD, Gotse Delchev
  - Medical centre Zdrave 1 OOD, Kozloduy
  - UMHAT Pulmed OOD - Pazardzhik, Department of Internal Diseases, Pazardzhik
  - MHAT Heart and Brain EAD, First department of Endocrinology and Metabolic Diseases, Pleven
  - MHAT Knyaginya Klementina - Sofia EAD, Sofia
  - MHAT Sveta Sofia EOOD, Department of Endocrinology and Metabolic diseases, Sofia
  - Acibadem City Clinic UMHAT Tokuda EAD, Endocrinology, Sofia
  - USHATE Akad. Ivan Penchev EAD, Second Clinic of Endocrinology, Sofia
  - Medical Institute of Ministry of interior, Sofia
  - Medical Centre - Clinic Nova EOOD, Varna
- Croatia (8):
  - Poliklinika Medikol Zagreb, Grad Zagreb
  - Opca bolnica Karlovac, Karlovac
  - Specijalna Bolnica za medicinsku rehabilitaciju Krapinske Toplice_Endocrinology, Krapinske Toplice
  - Poliklinika SLAVONIJA OSIJEK, Osijek
  - Clinical Hospital Centre Rijeka_Endocrinology, Rijeka
  - General Hospital Dr. Josip Bencevic_Diabetic department, Slavonski Brod
  - Opca bolnica Varazdin_Endocrinology, Varaždin
  - Poliklinika Solmed, Zagreb
- Germany (10):
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - Praxis am Markt Dr. Becker, Essen
  - MVZ im Altstadt-Carree Fulda GmbH - Zentrum für klinische Studien, Fulda
  - Diabetes-Zentrum-Wilhelmsburg GbR, Hamburg
  - Diabetologische Gemeinschaftspraxis Dr. Staudenmeyer und Dr. Schiwietz, Lingen
  - SMO.MD GmbH - Zentrum für klinische Studien, Magdeburg
  - Institut für Diabetesforschung Osnabrück, Osnabrück
  - ceda - Centrum für Diabetologie und Allgemeinmedizin Pohlheim, Pohlheim
  - Forschungszentrum Ruhr KliFoCenter GmbH, Kahrmann, Witten
- Hungary (5):
  - Debreceni Egyetem, Debrecen, Hajdú-Bihar
  - Komáromi Selye János Kórház, Komárom, Komárom-Esztergom
  - Óbudai Egészségügyi Centrum, Budapest, Pest County
  - Borbánya Praxis E.Ü. Kft., Nyíregyháza, Szabolcs-Szatmar Varmegye
  - Békés Vármegyei Központi Kórház, Gyula
- India (18):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - SSG Hospital, Baroda, Vadodara, Gujarat
  - Diacon Hospital Private Limited, Bangalore, Karnataka
  - Lifecare Hospital and Research Centre, Bengaluru, Karnataka
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - BSES MG hospital, Mumbai, Maharashtra
  - Shalini Tai Meghe Hospital and Research Center, Nagpur, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Arthur Asirvatham hospital,, Madurai, Tamil Nadu
  - NIZAM'S Institute of Medical Sciences, Hyderabad, Telangana
  - IPGME&R and SSKM Hospital, Kolkata, West Bengal
  - Rajiv Gandhi Centre for Diabetes and Endocrinology, J.N Medical College, Aligarh Muslim University, Aligarh
  - All India Institute of Medical Sciences (AIIMS), New Delhi
  - Jothydev's Diabetes & Research Center, Thriruvananthapuram
- Mexico (3):
  - Diseño y Planeación en Investigación Médica S.C., Guadalajara, Jalisco
  - Alliance CEINV Salud S.A. de C.V., Monterrey, Nuevo León
  - Centro de Estudios de Investigación Metabólicos y Cardio, Ciudad Madero, Tamaulipas
- Poland (20):
  - Gabinety Medyczne MATUSZEK Beata Matyjaszek-Matuszek Prywatna Praktyka Specjalistyczna, Lublin, Lesser Poland Voivodeship
  - EKAMED sp. z o.o., Lublin, Lublin Voivodeship
  - Przychodnie Grudziadz Sp. z o. o., Grudziądz, Mazovian Voivodeship
  - Legeartis Poradnie Specjalistyczne Sp. z o.o., Bialystok, Podlaskie Voivodeship
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok
  - NZOZ Vita-Diabetica Malgorzata Buraczyk, Bialystok
  - Centrum Kliniczno-Badawcze J.Brzezicki B.Gornikiewicz-Brzezicka Lekarze sp.p., Elblag
  - Specjalistyczny Gabinet Diabetologiczny Radoslaw Rumianowski, Gorzów Wielkopolski
  - SP ZOZ w Kalwarii Zebrzydowskiej, Kalwaria Zebrzydowska
  - Linden sp. z o.o. sp. k., Krakow
  - Diamond Clinic sp zoo, Krakow
  - Beata Miklaszewicz & Dariusz Dabrowski "CARDIAMED" s.j., Legnica
  - Serce Sp. z o.o., Leszno
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Centrum Terapii Wspolczesnej - J.M. Jasnorzewska S.K.A., Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej Przychodnia Specjalistyczna A Wittek H Rudzki Sp. j., Ruda Śląska
  - Lukmed 2 Sp. z o.o., Siedlce
  - Szpital Czerniakowski Sp. z o.o., Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Szyszko, Zabrze
  - Prywatna Praktyka Lekarska Anna Chudoba, Żyrardów
- Portugal (8):
  - Hospital de Cascais, Alcabideche
  - ULS Almada-Seixal E.P.E. - Hospital Garcia de Orta, Almada
  - ULS De Braga, E.P.E. - Hospital de Braga, Braga
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Hosp. das Forças Armadas_ Endocrinologia, Lisbon
  - Unidade Local de Saude de Sao Joao E.P.E, Porto
  - ULS De Matosinhos E.P.E.- Hospital Pedro Hispano, Senhora Da Hora, Matosinhos
  - Hospital Luz Arrabida, S.A., Vila Nova de Gaia
- Romania (8):
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - Poli Cardinal Med Srl, Reghin, Mureș County
  - CMI Dr. Pletea Noemi SRL, Bacau
  - SC Nutrilife SRL, Bucharest
  - Diabet Med SRL, Bucharest
  - Medical Practice SRL, Oradea
  - Spital Judetean De Urgenta Satu Mare, Satu Mare
  - Cabinet Medical Dr Geru SRL, Timișoara
- Thailand (5):
  - King Chulalongkorn Memorial Hospital_Endocrinology, Bangkok
  - Rajavithi Hospital_Diabetes and Endocrinology, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (7):
  - Başkent Üniversitesi Adana-Endokrinoloji, Adana /yüreği̇r
  - Ankara Bilkent Şehir Hastanesi-Dahiliye, Ankara
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi Hastanesi- Endokrinoloji, Battalgazi / Malatya
  - Göztepe Prof. Dr.Süleyman Yalçın Şehir Hastanesi- Dahiliye, Istanbul
  - Marmara Üniversitesi Pendik EAH- Endokrinoloji, Pendik/istanbul
  - Sivas Cumhuriyet Üniversitesi Hastanesi -Endokrinoloji, Sivas
  - Adana Şehir Eğitim ve Araştırma Hastanesi-Endokrinoloji, Yüreğir/Adana

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com